CLINICAL TRIAL: NCT03191188
Title: A Pilot Feasibility Trial of Thyroid Hormone Replacement in Dialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS#2014-1144; R03DK114642 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Thyroid Disease; Kidney Diseases, Chronic
MeSH Terms: conditions — Thyroid Diseases; Renal Insufficiency, Chronic | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levothyroxine (Experimental)
  Interventions: Drug: Levothyroxine Sodium
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Levothyroxine Sodium — Thyroid hormone supplement
  Arms: Levothyroxine
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo

SUMMARY:
Hypothyroidism, defined by elevated thyrotropin (TSH) levels, is a common endocrine complication of chronic kidney disease that has been associated with impaired quality of life and cardiovascular complications. While levothyroxine is one of the most frequently prescribed medications in chronic kidney disease patients, little is known about its efficacy and safety in this population. This study will investigate 1) whether levothyroxine adequately lowers thyrotropin (TSH) levels to therapeutic target ranges, and 2) if thyroid hormone replacement improves quality of life and cardiovascular markers, without leading to wasting in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent hemodialysis patients, elevated thyrotropin level, normal free thyroxine level.

Exclusion Criteria:

* Hyperthyroidism, active treatment with thyroid hormone replacement, prior thyroid malignancy, active pregnancy, active coronary ischemia or atrial fibrillation, osteoporosis, inability to provide consent without a proxy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Achievement of target TSH levels: serum TSH levels ranging from 0.5-3.0mIU/L | 12 weeks
  Number of patients achieving target TSH levels of 0.5-3.0mIU/L

SECONDARY OUTCOMES:
Health-related quality of life Short Form 36 questionnaire | Baseline and 12 weeks
  Change in Short Form 36 score
Serum Growth Differentiation Factor 15 (GDF15) level | Baseline and 12 weeks
  Change in GDF15 level
Serum soluble p-selectin level | Baseline and 12 weeks
  Change in soluble p-selectin level
Serum soluble CD40 ligand level | Baseline and 12 weeks
  Change in serum soluble CD40 ligand level
Body mass index | Baseline and 12 weeks
  Change in body mass index
Biceps skinfold | Baseline and 12 weeks
  Change in biceps skinfold
Triceps skinfold | Baseline and 12 weeks
  Change in triceps skinfold
Mid-arm circumference | Baseline and 12 weeks
  Change in mid-arm circumference
Mid-arm muscle circumference | Baseline and 12 weeks
  Change in mid-arm muscle circumference
Near infrared body fat percentage | Baseline and 12 weeks
  Change in near infrared body fat percentage
Subjective Global Assessment questionnaire | Baseline and 12 weeks
  Subjective Global Assessment questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Connie M. Rhee, MD, MSc, Principal Investigator — University of California, Irvine
Locations (1):
- University Dialysis Center of Orange, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhee CM, You AS, Nguyen DV, Brunelli SM, Budoff MJ, Streja E, Nakata T, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Thyroid Status and Mortality in a Prospective Hemodialysis Cohort. J Clin Endocrinol Metab. 2017 May 1;102(5):1568-1577. doi: 10.1210/jc.2016-3616. PMID 28324018
- [Background] Rhee CM, Kim S, Gillen DL, Oztan T, Wang J, Mehrotra R, Kuttykrishnan S, Nguyen DV, Brunelli SM, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Association of thyroid functional disease with mortality in a national cohort of incident hemodialysis patients. J Clin Endocrinol Metab. 2015 Apr;100(4):1386-95. doi: 10.1210/jc.2014-4311. Epub 2015 Jan 29. PMID 25632971
- [Background] Rhee CM, Ravel VA, Streja E, Mehrotra R, Kim S, Wang J, Nguyen DV, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Thyroid Functional Disease and Mortality in a National Peritoneal Dialysis Cohort. J Clin Endocrinol Metab. 2016 Nov;101(11):4054-4061. doi: 10.1210/jc.2016-1691. Epub 2016 Aug 15. PMID 27525529
- [Background] Rhee CM, Kalantar-Zadeh K, Streja E, Carrero JJ, Ma JZ, Lu JL, Kovesdy CP. The relationship between thyroid function and estimated glomerular filtration rate in patients with chronic kidney disease. Nephrol Dial Transplant. 2015 Feb;30(2):282-7. doi: 10.1093/ndt/gfu303. Epub 2014 Sep 21. PMID 25246335